CLINICAL TRIAL: NCT00903500
Title: Controlled Outcome Evaluations of a Daily Physical Activity Intervention for Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: BOF (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005/380
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daily physical activity
  Interventions: Behavioral: Daily physical activity, pedometer and counseling
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Daily physical activity, pedometer and counseling — Individual counseling session, telephone counseling (7 calls), given by a psychologist and a pedometer, based on cognitive behavioral therapy, the Diabetes Prevention Program, the first Step Program and Motivational Interviewing
  Arms: 1

SUMMARY:
The intervention consists of an individual counseling session, telephone counseling (7 calls), given by a psychologist, and a pedometer. The intervention is based on cognitive behavioral therapy, the Diabetes Prevention Program, the first Step Program and Motivational Interviewing. The taxonomy of behavior change techniques is also taken into account. The duration of the intervention is six months. The individual session takes place one week after the baseline measurements, together with the participants' follow-up appointment with their endocrinologist. The individual session takes place at the endocrinology department and is expected to last approximately 30 minutes. In addition to the session, the participants of the intervention group receive a pedometer and a pedometer diary for six months. Participants of the intervention group also receive telephone counseling from the psychologist during 24 weeks. They receive a call every two weeks for four weeks and then every four weeks for the next 20 weeks, good for a total of seven counseling calls. The calls are expected to last approximately 20 minutes. The Control Group has no intervention at all and receive their usual care.

ELIGIBILITY:
Inclusion Criteria:

* Minimum six months post-diagnosis of type 2 diabetes age between 35 and 75 years
* Treated by diet alone, oral hypoglycaemic medications, insulin or combination therapy
* No documented PA limitations
* Dutch speaking
* Having a telephone number

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Physical activity measured with an accelerometer, pedometer en the International Physical Activity Questionnaire (IPAQ) | At baseline, after the intervention (at 6 months) and one year after baseline
Health parameters: systolic and diastolic blood pressure, resting heart rate, waist circumference, weight, height | At baseline, after the intervention (at 6 months) and one year after baseline
Blood samples taken to determine:HBA1C, glucose, insulin, leptin, c-peptide, IGF-1, total cholesterol, HDL-c, LDL-C, triglycerides, APo-B, high sensitive C-reactive protein, vrij-t, DHEAS Oestradiol, Shbg, LH, FSH | At baseline, after the intervention (six months) and one year after baseline
Dexa scan | At baseline, after the intervention (six months) and one year after baseline

SECONDARY OUTCOMES:
Questionnaires on psycho-social determinants of physical activity, on environmental determinants of physical activity and a motivational questionnaire | At baseline, after the intervention and one year after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ilse De Bourdeaudhuij, Principal Investigator — University Ghent
Locations (1):
- Univerversity Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Van Dyck D, De Greef K, Deforche B, Ruige J, Tudor-Locke CE, Kaufman JM, Owen N, De Bourdeaudhuij I. Mediators of physical activity change in a behavioral modification program for type 2 diabetes patients. Int J Behav Nutr Phys Act. 2011 Sep 29;8:105. doi: 10.1186/1479-5868-8-105. PMID 21958233
- [Derived] De Greef K, Deforche B, Tudor-Locke C, De Bourdeaudhuij I. Increasing physical activity in Belgian type 2 diabetes patients: a three-arm randomized controlled trial. Int J Behav Med. 2011 Sep;18(3):188-98. doi: 10.1007/s12529-010-9124-7. PMID 21052886
- See also: Website of the University Ghent — http://www.ugent.be